CLINICAL TRIAL: NCT04207905
Title: Evaluation of the Healthy Michigan Plan Section 1115 Community Engagement Requirement Waiver
Status: Terminated | Type: Observational
Why Stopped: The Healthy Michigan Plan community engagement requirement was implemented on 1/1/2020. On 3/4/2020, a US District Court judge vacated the CMS approval of this policy, thereby suspending implementation of this RCT. This was not an IRB suspension.
Sponsor: University of Michigan (Other)
Collaborators: Michigan Department of Health and Human Services (Other)
Responsible Party: Principal Investigator, John Ayanian, Director, Institute for Healthcare Policy and Innovation, University of Michigan
Other Study IDs: HUM00168117
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Health Insurance
Keywords: Medicaid Expansion; Work Requirement; Community Engagement Requirement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exempt for Evaluation Purposes: Individuals who would have been subject to the Healthy Michigan Plan (HMP) work requirements but have been randomly assigned to a control group that is exempt from reporting for evaluation purposes
- Work Requirement: Individuals who are subject to the Healthy Michigan Plan (HMP) work requirements
  Interventions: Other: Healthy Michigan Plan (HMP) coverage with work requirements

INTERVENTIONS:
Other: Healthy Michigan Plan (HMP) coverage with work requirements — For those who are not in the Exempt for Research Purposes group, to be eligible for HMP coverage beginning January 1, 2020, enrollees ages 19-62 must report 80 hours per calendar month of community engagement activities, such as employment, education, job training, job search activities, participation in substance use disorder (SUD) treatment, or community service.
  Groups: Work Requirement

SUMMARY:
The Centers for Medicare & Medicaid Services (CMS) approved the renewal of the Healthy Michigan Plan (HMP) Section 1115 Demonstration Waiver on December 21, 2018, for the period January 1, 2019-December 31, 2023. This waiver provides approval for the state to require Medicaid expansion beneficiaries ages 19-62 to complete and report 80 hours per month of community engagement as a condition of eligibility, among other waiver provisions, beginning January 1, 2020. Community engagement activities include employment, education, job training, job search activities, participation in substance use disorder (SUD) treatment, or community service.

The State of Michigan will implement a randomized controlled trial (RCT) to evaluate the impact of community engagement requirements on Medicaid enrollment, health insurance coverage, self-reported health status, access to and utilization of health services, earnings, and employment, compared to a control group of HMP enrollees exempted from the community engagement requirement for purposes of the evaluation.

DETAILED DESCRIPTION:
Goals of the Demonstration

As stated by the Michigan Department of Health and Human Services (MDHHS), the overarching goals of the Healthy Michigan Plan (HMP) demonstration are to increase access to quality health care, encourage the utilization of high-value services, promote beneficiary adoption of healthy behaviors, and implement evidence-based practice initiatives.

The main objectives of MDHHS for HMP include:

* Improving access to healthcare for uninsured or underinsured low-income Michigan residents;
* Improving the quality of healthcare services delivered;
* Reducing uncompensated care;
* Strengthening beneficiary engagement and personal responsibility;
* Encouraging individuals to seek preventive care, adopt healthy behaviors, and make responsible decisions about their healthcare;
* Supporting coordinated strategies to address social determinants of health in order to promote positive health outcomes, greater independence, and improved quality of life;
* Helping uninsured or underinsured individuals manage their health care issues;
* Encouraging quality, continuity, and appropriate medical care.

The evaluation for this demonstration is focused on examining:

* The impact of the community engagement requirement on enrollees' employment, earnings and financial well-being; enrollment in other public support programs; health outcomes; and health insurance status (HMP, commercial health insurance, or uninsurance);
* The extent to which new eligibility and coverage policies impact:

  * Hospital uncompensated care
  * Insurance coverage in the state
  * Overall HMP enrollment and characteristics of HMP enrollees
  * Enrollees' health care utilization
  * Medicaid health service expenditures
* The impact HMP has had on enrollees' health outcomes, employment status, and financial well-being;
* The experiences of HMP enrollees who are disenrolled regarding insurance coverage status, access to care, and re-enrollment; and
* Medicaid program sustainability, including Medicaid expenditures.

The RCT design involves the random selection of a control group of HMP enrollees from across the state who are expected to be subject to the community engagement requirement but who are designated as being not subject to this requirement during the evaluation period (January 1, 2020 through December 31, 2023). This control group will be compared to an intervention group of HMP enrollees who will be subject to the community engagement requirement. Individuals who enroll in HMP after randomization occurs will not be eligible for inclusion in the control group.

The random selection of the control group (22,917 HMP enrollees, representing 10% of the individuals identified as subject to the work requirements as of November 2019) was performed in December 2019. This sample size for the control group will enable longitudinal analysis of key outcomes (e.g., employment, insurance coverage, self-reported health status, health services utilization, income, and credit outcomes) over the demonstration period, with sufficient statistical power to assess differences in these outcomes.

Data sources will include beneficiary surveys; state administrative data, including Medicaid enrollment files, Medicaid administrative claims, specialty behavioral health administrative claims, Michigan Care Improvement Registry immunization history, health risk assessment tables, cost-share tables, and other Medicaid tables; state workforce data, including state unemployment insurance program data; and public use data, including American Community Survey, Current Population Survey, Medicaid enrollment data from Medicaid Budget and Expenditure System (MBES), Medicaid and Medicare cost reports, Credit data, Behavioral Risk Factor Surveillance System, Healthcare Cost & Utilization Project (HCUP) inpatient discharge data, and program administrative cost data.

ELIGIBILITY:
Inclusion Criteria: Enrollees eligible for the HMP community engagement requirement, including:

* Adult HMP beneficiaries ages 19-62 who are not otherwise exempt.

Exclusion Criteria: Enrollees exempt from the community engagement requirement includiung:

* Pregnant women
* Primary caregivers of a family member under six years of age (limited to one caregiver per household)
* Caretakers of a dependent with a disability who needs full-time care (allowed for one beneficiary per household if there is only one dependent with a disability who meets the criteria specified above in the household)
* Caretakers of an incapacitated individual even if the incapacitated individual is not a dependent of the caretaker
* Beneficiaries considered medically frail
* Beneficiaries currently receiving temporary or permanent long-term disability benefits from a private insurer or from the government
* Beneficiaries diagnosed with an acute medical condition that would prevent them from complying with the requirements
* Beneficiaries who have been incarcerated within the last six months
* Beneficiaries currently receiving unemployment benefits from the state
* Beneficiaries under 21 years of age who had previously been in foster care placement in Michigan
* Full-time students.

Ages: 19 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy Michigan Plan enrollees subject to the community engagement requirement are eligible for the study. The RCT design involves the random selection by the State of Michigan or its designee of a control group of HMP enrollees from across the state who are expected to be subject to the community engagement requirement but who are designated as being not subject to this requirement during the evaluation period (January 1, 2020 through December 31, 2023). This control group will be compared to an intervention group of HMP enrollees who will be subject to the community engagement requirement. Individuals who enroll in HMP after randomization occurs will not be eligible for inclusion in the control group.
Sampling Method: Probability Sample
Enrollment: 892 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Insurance coverage | 3 years
  Insurance coverage (self-reported uninsurance, employer-sponsored insurance, other types of insurance)
Enrollment in Medicaid | 4 years
  Enrollment in Medicaid (Medicaid eligibility data)
Employment | 3 years
  Employment status (self-reported)
Employment record | 4 years
  Employment status (state unemployment insurance data)
Educational enrollment | 3 years
  Educational enrollment (self-reported)
Job training participation | 3 years
  Job training participation (self-reported)
Number of hours worked | 3 years
  Number of hours worked (self-reported)
Number of hours worked, recorded | 4 years
  Number of hours worked (state unemployment insurance data)
Earnings | 4 years
  Income (state unemployment insurance data)
Income | 4 years
  Income (Medicaid eligibility data)
Health status, overall | 3 years
  Health status, overall (self-reported)
Days poor physical health | 3 years
  Days poor physical health (self-reported)
Days poor mental health | 3 years
  Days poor mental health (self-reported)
Days limited in usual activities due to health | 3 years
  Days limited in usual activities due to health (self-reported)

SECONDARY OUTCOMES:
Emergency room (ER) visits | 4 years
  Emergency room (ER) visits in past 12 months (Medicaid claims and encounter data)
Hospital admissions in past 12 months | 4 years
  Hospital admissions in past 12 months (Medicaid claims and encounter data)
Financial well-being | 3 years
  Financial well-being (self-reported)
Material hardship | 3 years
  Material hardship (self-reported)
Credit report outcomes | 4 years
  Credit scores, debt past due, medical bills in collections, public records including evictions, bankruptcies, wage garnishments
Enrollment in TANF | 4 years
  Enrollment in Temporary Assistance for Needy Families (TANF enrollment data)
Enrollment in SNAP | 4 years
  Enrollment in Supplemental Nutrition Assistance Program (SNAP enrollment data)

CONTACTS AND LOCATIONS:
Overall Officials: John Z Ayanian, MD, MPP, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Healthy Michigan Plan evaluation webpage of the University of Michigan Institute for Healthcare Policy & Innovation — https://ihpi.umich.edu/signature-programs/healthy-michigan-plan-evaluation